CLINICAL TRIAL: NCT01166126
Title: Phase II Trial of mTOR Inhibitor Temsirolimus Combined With MEK Inhibitor AZD 6244 in Patients With BRAF Mutant Stage IV Melanoma
Brief Title: Temsirolimus/AZD 6244 for Treatment-naive With BRAF Mutant Unresectable Stage IV
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02846; NCI-2012-02846 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MCC-16066 (Other: H. Lee Moffitt Cancer Center and Research Institute); 8436 (Other: CTEP); P30CA076292 (NIH)
Record Dates: First submitted 2010-07-12; First posted 2010-07-20 (Estimated); Results first posted 2013-05-23 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2012-12

CONDITIONS: Mucosal Melanoma; Recurrent Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — temsirolimus; Sirolimus; AZD 6244

ARMS (1):
- Treatment (temsirolimus and selumetinib) (Experimental): Treatment Phase: This period begins with the first intravenous (through the vein) infusion of TEMSIROLIMUS and the first AZD6244 administration by mouth (visit 2, Week 1) and will continue until Week 8 (Visit 4).
  As many as 38 patients will receive the same dosage of TEMSIROLIMUS injected in the veins once a week for 8 weeks, and the AZD6244 will be given as capsules by mouth twice a day for 8 weeks. That is one cycle. The TEMSIROLIMUS and AZD6244 will be given to participants as an outpatient, unless admission to the hospital was needed for treatment of related side effects or underlying disease. The subsequent cycles of TEMSIROLIMUS and AZD6244 will be given every 8 weeks. The TEMSIROLIMUS will be injected in a vein over 30 minutes.
  The continuation phase begins with visits at weeks 12 in patients who receive at least two cycles of treatments.
  Interventions: Drug: temsirolimus; Drug: selumetinib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel
Drug: selumetinib — Given orally
  Other Names: ARRY-142886; AZD6244
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
The purpose of this study is to find out how often two investigational drugs that are given together will shrink the patient's tumor and how well they will prolong the time it takes their tumor to grow. The investigators also wish to find out how they affect certain substances in the patient's tumor and in their blood important for tumor growth. The combination of these drugs is experimental, and has not been proven to help treat melanoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the clinical response rate (Response Evaluation Criteria in Solid Tumors [RECIST]) and one-year overall survival to the study drugs temsirolimus and AZD6244 (selumetinib) hydrogen sulfate in BRAF V600E mutant unresectable stage IV melanoma.

SECONDARY OBJECTIVES:

I. Estimate 6-month progression-free survival in patients receiving temsirolimus and AZD6244 hydrogen sulfate.

II. Determine the pharmacodynamic effects of temsirolimus and AZD6244 on pERK, s6K, PTEN and mediators of apoptosis.

III. Determine the toxicity profile of temsirolimus with AZD6244 hydrogen sulfate.

OUTLINE:

Treatment Phase: This period begins with the first intravenous (through the vein) infusion of TEMSIROLIMUS and the first AZD6244 administration by mouth (visit 2, Week 1) and will continue until Week 8 (Visit 4).

As many as 38 patients will receive the same dosage of TEMSIROLIMUS injected in the veins once a week for 8 weeks, and the AZD6244 will be given as capsules by mouth twice a day for 8 weeks. That is one cycle. The TEMSIROLIMUS and AZD6244 will be given to participants as an outpatient, unless admission to the hospital was needed for treatment of related side effects or underlying disease. The subsequent cycles of TEMSIROLIMUS and AZD6244 will be given every 8 weeks. The TEMSIROLIMUS will be injected in a vein over 30 minutes.

The continuation phase begins with visits at weeks 12 in patients who receive at least two cycles of treatments.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have read, understood, and provided written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization after the nature of the study has been fully explained
* Subjects with a histologic diagnosis of unresectable stage IV melanoma (may include mucosal melanoma)
* Tumor must be BRAF V600E mutation positive from a certified lab
* At least 4 weeks since any previous treatment (surgery, radiotherapy, or systemic treatment)
* Women should be either: post-menopausal for at least 1 year; surgically incapable of bearing children; or utilizing a reliable form of contraception during the study and for at least 4 months after the final study drug infusion or ingestion; women of childbearing potential must have a negative serum hCG-beta pregnancy test conducted during the screening period
* Men who may father a child must agree to the use of male contraception for the duration of their participation in the trial and for at least 4 months after the final temsirolimus and AZD6244 hydrogen sulfate administration
* Life expectancy >= 3 months
* ECOG performance status of 0 or 1
* Patients with brain metastases treated with surgery, radiation, or stereotactic radiosurgery who are without evidence of progression in their brain metastases after MRI imaging performed at least 30 days after treatment, and are not taking systemic steroids will be eligible
* WBC >= 3000 cells/mm^3
* ANC >= 1500 cells/mm^3
* Platelets >= 100,000/mm^3
* Hematocrit >= 30%
* Hemoglobin >= 9 g/dL
* Creatinine =< 2.0 mg/dL
* AST/ALT =< 2 x ULN
* Bilirubin =< 1.5 x ULN, (except subjects with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dL)
* HIV negative
* HBsAg negative
* Anti-HCV Ab nonreactive; if reactive, subject must have a negative HCV RNA qualitative PCR
* Patients with hyperlipidemia must have adequate control with a lipid lowering agent

Exclusion Criteria:

* Any prior malignancy except for the following: adequately treated basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix, or any other cancer from which the subject has been disease-free for at least 5 years
* Active infection, requiring therapy, chronic active HBV or HCV; patients with HIV, who have adequate CD4 counts and who do not require HAART therapy, are NOT excluded
* Pregnancy or nursing: due to the possibility that temsirolimus and AZD6244 hydrogen sulfate could have a detrimental effect on the developing fetus or infant, exposure in utero or via breast milk will not be allowed
* Any underlying medical condition which, in the opinion of the principal investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events
* Prior treatment with temsirolimus or AZD6244 or any prior mTOR or MEK inhibitor
* Evidence or history of significant cardiac, pulmonary, hepatic, renal, psychiatric or gastrointestinal disease that would make the administration of temsirolimus or AZD6244 hydrogen sulfate unsafe
* Tumor that is BRAF V600E mutation negative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ragini Kudchadkar, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Up to 35 subjects with a histologic diagnosis of unresectable Stage IV melanoma were to be enrolled into this study over 24 months.
Pre-assignment Details: 11 of 15 patients consented were not eligible to receive the study drug after screening.
Groups:
- Treatment (Temsirolimus and Selumetinib): Treatment Phase: This period begins with the first intravenous (through the vein) infusion of TEMSIROLIMUS and the first AZD6244 administration by mouth (visit 2, Week 1) and will continue until Week 8 (Visit 4).
  Investigators planned for as many as 38 patients to receive the same dosage of TEMSIROLIMUS injected in the veins once a week for 8 weeks, and the AZD6244 would be given as capsules by mouth twice a day for 8 weeks. That is one cycle. The TEMSIROLIMUS and AZD6244 would be given to participants as an outpatient, unless admission to the hospital was needed for treatment of related side effects or underlying disease. The subsequent cycles of TEMSIROLIMUS and AZD6244 would be given every 8 weeks. The TEMSIROLIMUS would be injected in a vein over 30 minutes.
  The continuation phase would begin with visits at weeks 12 in patients who received at least two cycles of treatments.
Period: Overall Study
Arm/Group | Treatment (Temsirolimus and Selumetinib)
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All baseline participants
Arm/Group | Treatment (Temsirolimus and Selumetinib)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 52.5 [39 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response (CR) and Partial Response (PR)
Description: Anti-tumor response (CR+PR) was defined by Response Evaluation Criteria in Solid Tumors (RECIST).
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: 1 year
Population: All participants
Measure: Number; unit: participants
Groups:
- Treatment (Temsirolimus and Selumetinib): Treatment Phase: This period began with the first intravenous (through the vein) infusion of TEMSIROLIMUS and the first AZD6244 administration by mouth (visit 2, Week 1) and will continue until Week 8 (Visit 4).
  Investigators planned for as many as 38 patients to receive the same dosage of TEMSIROLIMUS injected in the veins once a week for 8 weeks, and the AZD6244 would be given as capsules by mouth twice a day for 8 weeks. That is one cycle. The TEMSIROLIMUS and AZD6244 would be given to participants as an outpatient, unless admission to the hospital was needed for treatment of related side effects or underlying disease. The subsequent cycles of TEMSIROLIMUS and AZD6244 would be given every 8 weeks. The TEMSIROLIMUS would be injected in a vein over 30 minutes.
  The continuation phase would begin with visits at weeks 12 in patients who received at least two cycles of treatments.
Arm/Group | Treatment (Temsirolimus and Selumetinib)
Number analyzed (Participants) | 4
participants
  Complete Response | 0
  Partial Response | 0

2. Primary Outcome: Number of Participants With Overall Survival (OS) at One Year
Description: The one-year overall survival of the combination of temsirolimus and AZD6244 Hydrogen Sulfate.
Time Frame: 1 year post last treatment
Measure: Number; unit: participants
Arm/Group | Treatment (Temsirolimus and Selumetinib)
Number analyzed (Participants) | 4
participants | 0

3. Secondary Outcome: Number of Participants With Progression Free Survival (PFS) at 6 Months.
Description: Patients will be evaluated by physical examination and imaging assessments (brain MRI and CT scans of the chest, abdomen and pelvis). Disease progression will be defined by RECIST criteria on physical exam or diagnostic imaging assessments that are attributed to metastatic melanoma.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: 6 months from day 1 of treatment
Measure: Number; unit: participants
Arm/Group | Treatment (Temsirolimus and Selumetinib)
Number analyzed (Participants) | 4
participants | 1

4. Secondary Outcome: Number of Participants With Related Serious Adverse Events (SAEs)
Description: Toxicities assessed using NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v4.0.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Treatment (Temsirolimus and Selumetinib)
Number analyzed (Participants) | 4
participants | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment (Temsirolimus and Selumetinib)
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Temsirolimus and Selumetinib) (N=4)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Neoplasms benigh, malignant and unspecified (incl cysts and polyps) - other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Temsirolimus and Selumetinib) (N=4)
Constipation (Gastrointestinal disorders) | 4 (4)
Mucositis oral (Gastrointestinal disorders) | 4 (20)
Nausea (Gastrointestinal disorders) | 3 (8)
Diarrhea (Gastrointestinal disorders) | 2 (6)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - other (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Fatigue (General disorders) | 4 (8)
Fever (General disorders) | 3 (5)
Edima - limbs (General disorders) | 2 (3)
Pain (General disorders) | 2 (4)
Chills (General disorders) | 1 (1)
Edema - face (General disorders) | 1 (1)
General disorders and administration site conditions - other (General disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Paresthesia (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (3)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Lipase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Cholesterol high (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (14)
Serum amylase increased (Investigations) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (5)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Blood and lymphatic system disorders - other (Blood and lymphatic system disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 1 (1)
Hepatobiliary disorders - other (Hepatobiliary disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
The study was terminated due to overall low accrual and a high rate of screening failures. Accrual goal was 38 participants and only 4 participants were actually treated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less